CLINICAL TRIAL: NCT00454454
Title: Display Enhanced TEsting for Cognitive Impairment and Traumatic Brain Injury
Brief Title: Virtual Reality Helmet to Test for Problems With Memory
Acronym: DETECT
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Wallace H. Coulter Foundation (Other)
Responsible Party: Principal Investigator, David Wright, Associate Professor, Emory University
Other Study IDs: 797-2002
Record Dates: First submitted 2007-03-28; First posted 2007-03-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Memory
Keywords: memory; display enhanced testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
The purpose of this research study is to compare a virtual reality display device with the standard neuropsychological evaluation for detecting mild cognitive impairment (problems with memory, concentration, reaction time, etc.).

DETAILED DESCRIPTION:
Since many individuals with mild cognitive impairment (MCI) appear to function normally, MCI may often be recognizable through testing in advance of any changes noticed by family members or caregivers. Early and frequent testing can therefore trigger an earlier diagnosis, which may increase the effectiveness of currently available medications used to delay onset of Alzheimer's symptoms. Primary care and geriatric physicians currently lack the necessary tools required for quick and accurate MCI screening in the doctor's office environment. The current industry-standard is a battery of pen & paper neuropsychological tests that require 1.5 hours in a quiet room with a neuropsychologist.

Comparison: virtual reality display device compared to the standard neuropsychological evaluation for detecting mild cognitive impairment (problems with memory, concentration, reaction time, etc.).

ELIGIBILITY:
Inclusion Criteria:

* 65 yrs of age and older
* MMSE of 18 or greater or mini-cog of 4 or greater
* Ability to read
* Informed consent given

Exclusion Criteria:

* Visual, hearing or physical impairment that would limit ability to use the virtual reality helmet or control device
* Non-English speaking

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: geriatric clinic, retirement facilities
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2007-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Wright, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Wesley Woods Health Center, Atlanta, Georgia
  - Wesley Woods Outpatient Clinic, Atlanta, Georgia

REFERENCES:
- [Result] Wright DW, Nevarez H, Kilgo P, LaPlaca M, Robinson A, Fowler S, Brumfield J, Goldstein FC. A novel technology to screen for cognitive impairment in the elderly. Am J Alzheimers Dis Other Demen. 2011 Sep;26(6):484-91. doi: 10.1177/1533317511426133. Epub 2011 Nov 22. PMID 22110158